CLINICAL TRIAL: NCT03740841
Title: Evaluation of the Effects of LUNII on Pre-operative Anxiety and on the Post-operative Period in Children With Cleft Lip and Palate Admitted for Alveolar Bone Graft: Pilot Study
Acronym: LUNII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K180306J; 2018-A00758-47 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-03

CONDITIONS: Cleft Lip and Palate
Keywords: Per-operative stress; per-operative anxiety; pediatric surgery
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUNII (Other): The interactive story teller LUNII is delivered to the child the day before surgery, during the usual pre-operative medical visit.
  Interventions: Behavioral: Interactive story teller LUNII
- Without LUNII (No Intervention): Usual pre-operative visit.

INTERVENTIONS:
Behavioral: Interactive story teller LUNII — Use of the interactive story teller LUNII by the child from the pre-operative visit to the discharge.
  Arms: LUNII

SUMMARY:
The literature on the effects of various devices on per-operative anxiety is scarce. There is currently no study on the effects of an interactive storyteller on per-operative anxiety in pediatric surgery.

The interactive story teller LUNII (available over the counter in France) would reduce pre-operative anxiety, with post-operative effects on pain and hospitalization time.

DETAILED DESCRIPTION:
The literature on the effects of various devices on per-operative anxiety is scarce. There is currently no study on the effects of an interactive storyteller on per-operative anxiety in pediatric surgery.

The interactive story teller LUNII (available over the counter in France) would reduce pre-operative anxiety, with post-operative effects on pain and hospitalization time.

Patients admitted for an alveolar bone graft with an iliac donor site as part of the treatment of their cleft lip and palate will be include for two reasons:

1. It is a homogeneous population - same condition, same treatment, same age at surgery, standardized procedure;
2. It is a population with long individual medical histories and, potentially, subjected to significant surgery-related stress.

Patients will be randomized into two groups: with LUNII and without LUNII.

In the LUNII group, the interactive story teller LUNII will be delivered the day before surgery during the pre-operative medical visit.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 6 years.
* Alveolar bone graft with iliac crest donor site in children with unilateral or bilateral cleft lip and palate
* Primary alveolar bone graft or first side when bilateral cleft
* Followed at Necker since birth and operated according to the protocol used in the department.
* Consent signed by the holder (or holders) of parental authority

Exclusion Criteria:

* Medical care different from the usual protocol applied in the service (secondary surgery, age > 7 years)
* Known psychomotor delay, associated rare syndrome or disease, known psychiatric disorders, other surgical procedures between hard palate closure and alveolar bone graft
* Possession and/or prior use of LUNII by the child

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Yale Preoperative Anxiety Scale (mYPAS ) | At the entrance into the operating room
  Questionnaire, completed in the operating room by an independent observer preferably without knowledge about the child, made of 22 items divided into 5 categories. The score ranges from 5 (minimum anxiety) to 20 (maximum anxiety)
Yale Preoperative Anxiety Scale (mYPAS ) | At the time of anesthetic induction
  Questionnaire, completed in the operating room by an independent observer preferably without knowledge about the child, made of 22 items divided into 5 categories. The score ranges from 5 (minimum anxiety) to 20 (maximum anxiety)
Number of hours spent with the interactive story teller LUNII before surgery | Day of surgery (D0)
  Number of hours spent with the interactive story teller LUNII

SECONDARY OUTCOMES:
Analgesic administration | Up to 1 week
  Evaluation of analgesic administration after surgery during hospital stay
Visual Analogue pain Scale (EVA) | Up to 1 week
  Self-assessment of pain by a graduated ruler of 0 (no pain) at 100 millimeters (maximum pain imaginable), twice a day during hospitalization
Duration between the operation and the first survey | Up to 1 week
  Duration between the operation and the first survey
Length of hospitalization | Up to 1 week
  Length of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hossein Khonsari, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No